CLINICAL TRIAL: NCT01730079
Title: Near Infra-Red Spectroscopy (NIRS) in Neurodevelopmental Disorders and Typically Developing Children
Brief Title: Near Infrared Spectroscopy in Children With Autism and ADHD
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130007; 13-M-0007
Record Dates: First submitted 2012-11-17; First posted 2012-11-21 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2017-04-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Attention Deficit Disorder; Attention Deficit Hyperactivity Disorder; Autism; Autism Spectrum Disorders
Keywords: Attention Deficit Hyperactivity Disorder; Autism; Near Infrared Spectroscopy; Brain Activity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Near-infrared spectroscopy (NIRS) is a functional imaging technique that can be uses light to study brain function while allowing for movement. To look at blood flow in the brain, NIRS uses a low-power light source with detectors that see how the light changes as it passes through brain tissue. Brain blood flow can indicate which parts of the brain are active during different tasks. Researchers want to study children with attention deficit hyperactivity disorder (ADHD) and autism spectrum disorders (ASD) and will use NIRS to compare the blood flow in the brain of children with ADHD and ASD with that of typically developing children.

Objectives:

* To see how well NIRS can detect changes in brain blood flow during tests of thinking and memory in children.
* To compare blood flow in the brains of typically developing children and those with ADHD or ASD.

Eligibility:

- Children between 4 and 8 years of age with ASD, ADHD, or children with no psychiatric diagnoses.

Design:

* Participants will be screened for eligibility. Those who are taking stimulant medication for ADHD or ASD will need to stop taking it for 3 days before the study visit.
* After participating in a screening assessment, all participants will have one study visit. At this visit, they will have be asked to complete two tasks during a NIRS scan. For both tasks, they will react to images on a computer screen. This visit will last about 2 hours.
* This is a testing study only. No blood or other samples will be needed for this study.

DETAILED DESCRIPTION:
Objective: to test whether Near Infra-Red Spectroscopy (NIRS) can be used to monitor cognitive brain function and detect markers for differentiation of Autism Spectrum Disorders (ASD) and Attention Deficit Hyperactivity Disorder (ADHD).

Study population: Children with ASD, ADHD, and typically developing children, all between 4 and 8 years of age.

Design: The study will investigate NIRS signal changes while children with ASD, ADHD, and typically developing children perform well-known functional tasks.

Outcome Measures: Graded changes in blood flow and oxygen, measured with NIRS, in response to different functional tasks.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children will be between 4 to 8 years of age (4 years, 0 months to 8 years, 11 months). English speakers only will be recruited for the study, because the language measures/tests and stimuli being used are in English and were developed and standardized on English-only samples.

Typically Developing Group:

-Development in nonverbal and verbal areas within age expectations (per scores onthe Differential Ability Scales, Second Edition or the Wechsler Preschool and Primary Scale of Intelligence Fourth Edition , no more than 1.5 standard deviation below the mean)

ASD Group:

-Diagnosis of Autistic Disorder, Asperger s disorder, or Pervasive Developmental Disorder - Not Otherwise Specified (PDD NOS), based on diagnostic evaluation conducted through a separate screening protocol

ADHD Group:

-Diagnosis of ADHD based on diagnostic evaluation conducted through a separate screening protocol Minimum Nonverbal IQ of 80; Minimum Verbal IQ score of 60

EXCLUSION CRITERIA:

All children who meet the following criteria:

* Primary language spoken at home is other than English
* Any skin disease that affects the scalp
* Past or present vascular disease, such as lupus, ankylosing spondylitis or scleroderma.
* Known adverse reaction to latex
* Presence or history of medical conditions known to affect cerebral anatomy, such as known cysts, arterivenous malformations or cortical tubers.
* Head trauma with loss of consciousness lasting longer than 5 seconds in the last year or any evidence of functional impairment due to and persisting after head trauma
* Motor movement disorder which may cause sudden excessive movement, such as Tourette s disorder
* Birth before 32 weeks of gestation. Premature birth can have a profound effect on brain function and structure
* A known neurological or neurogenetic condition affecting the central nervous system, such as epilepsy, cerebral palsy, neurofibromatosis, velo-cardiofacial syndrome.
* Color blindness

Typically Developing Group:

* Cognitive impairment, defined as Nonverbal IQ below 80, or signs of ASD or ADHD
* Confirmed diagnosis of any DSM-IV-TR Axis I disorder
* Taking medications for neuropsychiatric disorders such as antidepressants, antipsychotics, mood stabilizers, anxiolytics or any medication used to treat ADHD (psychostimulants, atomoxetine (Strattera ), bupropion (Wellbutrin ), tricyclic antidepressants (like impramine), clonidine, guanfacine, or modafinil (Provigil ).

ASD Group:

* Taking medications for neuropsychiatric disorders: such as antidepressants, antipsychotics, mood stabilizers, or anxiolytics. Some medications used to treatment for ADHD are also exclusionary for all children - including atomoxetine (Strattera ), bupropion (Wellbutrin ), tricyclic antidepressants (like impramine), clonidine, guanfacine, or modafinil (Provigil ). Children with ASD who take stimulants (like Ritalin, adderall, concerta and vyvanse) may be able to participate if they are willing and able to stop stimulant medications for 2 days on 1 occasion for the study
* A known neurological or neurogenetic condition affecting the central nervous system, such as epilepsy, cerebral palsy, neurofibromatosis, velo-cardiofacial syndrome.

ADHD Group:

* Taking medications for neuropsychiatric disorders: such as antidepressants, antipsychotics, mood stabilizers, or anxiolytics. Some medications used to treatment for ADHD are also exclusionary for all children - including atomoxetine (Strattera ), bupropion (Wellbutrin ), tricyclic antidepressants (like impramine), clonidine, guanfacine, or modafinil (Provigil ). Children with ASD who take stimulants (like Ritalin, adderall, concerta and vyvanse) may be able to participate if they are willing and able to stop stimulant medications for 2 days on 1 occasion for the study
* Other psychiatric diagnoses (including ASD, anxiety and depression), except for comorbid oppostional defiant disorder

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2012-10-23; Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Graded changes in blood flow and oxygen, measured with NIRS, in response to different functional tasks.

SECONDARY OUTCOMES:
Differential activity according to region of the frontal cortext and task elements.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey E Thurm, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boas DA, Dale AM, Franceschini MA. Diffuse optical imaging of brain activation: approaches to optimizing image sensitivity, resolution, and accuracy. Neuroimage. 2004;23 Suppl 1:S275-88. doi: 10.1016/j.neuroimage.2004.07.011. PMID 15501097
- [Background] Carlsson J, Lagercrantz H, Olson L, Printz G, Bartocci M. Activation of the right fronto-temporal cortex during maternal facial recognition in young infants. Acta Paediatr. 2008 Sep;97(9):1221-5. doi: 10.1111/j.1651-2227.2008.00886.x. PMID 18627358
- [Background] Elwell CE, Henty JR, Leung TS, Austin T, Meek JH, Delpy DT, Wyatt JS. Measurement of CMRO2 in neonates undergoing intensive care using near infrared spectroscopy. Adv Exp Med Biol. 2005;566:263-8. doi: 10.1007/0-387-26206-7_35. PMID 16594161